CLINICAL TRIAL: NCT06978335
Title: Acupoint Stimulation Intervention Improves Postoperative Wound Pain and Mobility in Patients With Abdominal Surgery
Brief Title: Acupoint Stimulation Improves Postoperative Wound Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: (1090)113A-20
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Surgeries; Pain; Acupuncture Points
Keywords: acupoint stimulation; postoperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Acupoint Stimulation (Experimental): Acupoint stimulation was administered on six points and auricular points on three points on the left ear, additional auricular points were selected according to the abdominal organ involved in surgery and its corresponding meridian representation on the auricle.
  Interventions: Other: Acupoint Stimulation
- Control: Sham Acupoint Stimulation (Sham Comparator)
  Interventions: Other: Sham Acupoint Stimulation

INTERVENTIONS:
Other: Acupoint Stimulation — This intervention involves acupoint stimulation and auricular acupressure. Stimulation of selected body acupoints is administered by trained personnel following a standardized protocol. The intervention is provided once daily for three consecutive days, beginning post-surgery. For auricular acupressure, additional auricular points are chosen based on the involved abdominal organ and its corresponding viscera-meridian locations on the auricle. Vaccaria seeds are applied to the selected points with adhesive patches, and patients are instructed to apply pressure to the points regularly throughout the day.
  Arms: Experimental: Acupoint Stimulation
Other: Sham Acupoint Stimulation — Participants in this group will receive a sham acupoint stimulation procedure. Acupoint stimulation will be using identical procedures to the experimental group, without applying pressure. No stimulation or manipulation was performed. The frequency and timing of the sham intervention matched that of the experimental group.
  Arms: Control: Sham Acupoint Stimulation

SUMMARY:
Postoperative pain remains one of the most common and distressing symptoms experienced by surgical patients. Poorly managed postoperative pain can impede recovery, reduce patient willingness to mobilize, increase the risk of complications, and negatively affect overall quality of life. Currently, opioids and nonsteroidal anti-inflammatory drugs (NSAIDs) are the primary pharmacological strategies for managing postoperative pain. However, these medications often carry the risk of adverse effects and may not adequately address all aspects of patient comfort and recovery.

In response to this challenge, this study aims to evaluate the effects of a non-pharmacological, non-invasive intervention-acupoint stimulation-on postoperative wound pain and mobilization in patients undergoing abdominal surgery. Ultimately, this study seeks to contribute to the development of more diversified and patient-centered pain management strategies, with the expectation that the integration of Chinese and Western medicine will lead to improved patient care and enhanced postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Surgical wound length ≥ 10 cm
* American Society of Anesthesiologists (ASA) physical status classification I to III
* Receiving intravenous patient-controlled analgesia (IV PCA)
* Clear consciousness and ability to communicate
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Presence of arrhythmia
* Implanted artificial cardiac pacemaker
* Cutaneous lesions at the acupoint or auricular application sites
* History of chronic pain or abdominal surgery within the past 6 months
* Non-ambulatory status prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measured by Visual Analog Scale (VAS) | At 1, 4, 12, 24, 48, and 72 hours post-surgery
  Pain intensity will be assessed using the Visual Analog Scale (VAS). The primary analysis will focus on changes in pain intensity over time between the two groups.

SECONDARY OUTCOMES:
Pain Impact Assessed by Brief Pain Inventory - Taiwan Version (BPI-Taiwan) | On postoperative Day 3
  The Brief Pain Inventory - Taiwan version (BPI-Taiwan) will be used to assess the impact of pain on various aspects of daily functioning. Total and subscale scores will be analyzed to evaluate differences in pain interference between the two groups.

OTHER OUTCOMES:
Total Analgesic Consumption Within 72 Hours After Surgery | Within 72 hours after surgery
  This outcome evaluates whether acupoint stimulation reduces the need for postoperative analgesics.
Time to First Ambulation After Surgery | Within 72 hours after surgery
  Time from completion of surgery to the first successful ambulation will be recorded. Recorded as an indicator of overall postoperative mobility and functional recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Hsin General Hospital, Taipei, Peitou Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No